CLINICAL TRIAL: NCT03794635
Title: A Communication-Based Intervention for Cancer Patient-Caregiver Dyads to Increase Engagement Treatment Planning and Reduce Caregiver Burden
Brief Title: An Intervention to Help Patients and Caregivers Manage Stress and Improve Communication Skills When Talking About Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-530
Record Dates: First submitted 2018-12-21; First posted 2019-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Cancer; Locally Advanced Cancer; Thoracic Cancer; Gynecologic Cancer; Genitourinary Cancer; Lymphoma
Keywords: Latina; Latino; Spanish; Caregiver; 18-530; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Neoplasm Metastasis; Urogenital Neoplasms; Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): Latino/a advanced cancer patients
  Interventions: Behavioral: Weekly 45 minute Sessions
- Caregivers (Experimental): Caregivers of Latino/a advanced cancer patients
  Interventions: Behavioral: Weekly 45 minute Sessions

INTERVENTIONS:
Behavioral: Weekly 45 minute Sessions — The current intervention consists of seven, weekly,45-minute sessions conducted over the telephone using the TAC manual workbook. MSK-approved platforms (such as Webex or Cisco Jabber) can be used for telephone calls in this study. There will be two versions of the intervention used for this study:
  1. A culturally tailored version for Latinx participants refined during Phase 1 of this study (available in English and Spanish)
  2. A version of the intervention that was not culturally tailored for Latinx patients and caregivers developed in previous work. The two interventions differ in minor content areas. The culturally tailored intervention for Latinx participants and the non-tailored intervention for non-Latinx participants will be used. Interventions will occur weekly with a plus three-week window.
  Characteristics of prognostic discussions between patients and caregivers and health providers will be assessed at baseline and post-intervention.

SUMMARY:
This study will test an intervention to improve patients' and their caregivers' ability to manage difficult emotions and communicate about the patient's illness. There will be two versions of the intervention used for this study: a culturally tailored version for Latinx participants refined during Phase 1 of this study, and a version of the intervention that was not culturally tailored for Latinx patients and caregivers developed in previous work. The two interventions differ in minor content areas. We will use the culturally tailored intervention for Latinx participants and the non-tailored intervention for non-Latinx participants. This culturally sensitive intervention has the potential to reduce Latino/a patient and caregiver distress and improve patient and caregiver quality of life, shared understanding of the patient's illness, and patients' and caregivers' ability to discuss, identify, and document patients' treatment preferences. The intervention is designed to minimize burden to patients, caregivers, and healthcare institutions to allow for easy integration into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

For Patients:

* Self-identifies as Latino/a
* Diagnosis of poor prognosis advanced cancer defined as: (1) locally advanced or metastatic cancer (i.e., thoracic, gynecological, genitourinary cancer, pancreatic or lymphoma) or (2) disease progression following at least first line treatment
* Fluent in English or Spanish
* Age 18 or older
* Has a primary informal caregiver (as defined by an unpaid individual who provides the patient with emotional, physical, and/or practical support) who is willing and able to participate in the study
* Score of </= 10 on the Blessed Orientation-Memory-Concentration Test (BOMC)
* To assess whether a prognostic discussion occurred, the oncologist must answer "Yes" to the following: "Have you discussed the any of the following with Mr./Mrs./Ms. [INSERT PATIENT"S NAME]: If his/her cancer is curable, if his/her cancer is terminal, or his/her life expectancy: Yes/No Note: This question will be included in the email in which study staff request permission to contact the patient.
* As per self-report, residency in New York or ability to complete sessions in New York to ensure that provision of TAC is covered by the professional licenses of TAC interventionists (i.e., social workers licensed in New York State) - AIMS 2 and 3 ONLY
* Able to communicate over the phone for sessions
* Willingness to be audio-recorded for assessments and study sessions

For Caregivers:

* Is a primary informal caregiver (as defined by an unpaid individual who provides the patient with emotional, physical, and/or practical support) for a MSK patient
* Fluent in English or Spanish
* Age 18 or older
* Score of </= 10 on the Blessed Orientation-Memory-Concentration Test (BOMC)
* As per self-report, residency in New York or ability to complete sessions in New York to ensure that provision of TAC is covered by the professional licenses of TAC interventionists (i.e., social workers licensed in New York State) - AIMS 2 and 3 ONLY
* Able to communicate over the phone for sessions
* Willingness to be audio-recorded for assessments and study sessions

Psychosocial expert eligibility requirements:

* Current clinical practice and/or research with advanced cancer patients
* A history of 5+ years working with advanced cancer patients. Experts across disciplines (e.g., social work, psychology) may be enrolled.
* Fluent in English as self-reported by a fluency of "Very well"

Exclusion Criteria:

For Patients

* As judged by the consenting professional, treating physician or self-report, too weak or cognitively impaired to participate in the intervention and complete the assessments
* Receiving hospice at the time of enrollment
* Deemed inappropriate for the study by their treating physician
* As per medical record or self-report, currently being treated for schizophrenia, substance use or dependence, and/or bi-polar disorder

For Caregivers:

* As judged by the consenting professional, treating physician or self-report, too weak or cognitively impaired to participate in the intervention and complete the assessments
* As per self-report, currently being treated for schizophrenia, substance use or dependence, and/or bi-polar disorder

Patient-Caregiver Dyads:

* Both dyad members respond "b" or "d" on the item in Appendix K, "How would you describe your/the patient"s health status: a) Relatively healthy, b) Relatively healthy and terminally ill, c) Seriously ill but not terminally ill, or d) Seriously and terminally ill" and respond "months" on the item "When you think about your/the patient's life expectancy, do you think in terms of months or years."

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of patient-caregiver communication-based intervention defined by participant enrollment | 3 months
Feasibility of patient-caregiver communication-based intervention defined by participant retention | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Trevino, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org